CLINICAL TRIAL: NCT04303559
Title: Multicenter, Randomized Phase III Inhibitor Prevention Trial, Comparing Eloctate vs. Emicizumab to Prevent Inhibitor Formation in Severe Hemophilia A
Brief Title: The Hemophilia Inhibitor Prevention Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The INHIBIT Trials IDSMB, in a letter dated 05-18-22, recommended, given the slow enrollment, that the INHIBIT Trials be discontinued due to futility.
Sponsor: Margaret Ragni (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Margaret Ragni, Professor of Medicine and Clinical and Translational Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO19040140; H30MC24050 (Other Grant/Funding Number: (HRSA) Health Resources and Services Administration)
Record Dates: First submitted 2020-03-02; First posted 2020-03-11 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia A Without Inhibitor
Keywords: hemophilia A; eloctate; Emicizumab; inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein; emicizumab

STUDY DESIGN:
Intervention Model Description: This is a phase III open-label, randomized controlled trial comparing two drugs in the prevention of hemophilia inhibitor formation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eloctate (Active Comparator): Arm A: Eloctate 65 IU/kg will be administered weekly by intravenous infusion in previously untreated children with severe hemophilia A beginning before the first bleed and continued up to 48 weeks.
  Interventions: Drug: Eloctate Injectable Product
- Emicizumab (Experimental): Arm B: Emicizumab 1.5 mg/kg will be administered weekly by subcutaneous injection (following 3 mg/kg/wk x4 induction) in previously untreated children with severe hemophilia A beginning before the first bleed and continue up to 48 weeks.
  Interventions: Drug: Emicizumab Injection [Hemlibra]

INTERVENTIONS:
Drug: Eloctate Injectable Product — This is a factor VIII-Fc fusion protein.
  Other Names: rFVIIIFc
  Arms: Eloctate
Drug: Emicizumab Injection [Hemlibra] — This is a bispecific monoclonal antibody FVIII mimic.
  Other Names: Hemlibra
  Arms: Emicizumab

SUMMARY:
This is a multi-center randomized phase III clinical trial, the Inhibitor Prevention Trial, in which Eloctate will be compared with Emicizumab, using adaptive design, to prevent inhibitors in patients with severe hemophilia A.

DETAILED DESCRIPTION:
This is a multi-center randomized phase III clinical trial, the Inhibitor Prevention Trial, in which consecutive hemostatic agents will be compared using adaptive design to prevent inhibitors in patients with severe hemophilia A. This adaptive design is necessary as randomized trials in rare diseases are otherwise not possible. This adaptive design is necessary as randomized trials in rare diseases are otherwise not possible. The INHIBIT Clinical Trials Platform includes two linked trials, the Inhibitor Prevention Trial (Prevention Trial) and the Inhibitor Eradication Trial (Eradication Trial) that will be conducted at up to 41 U.S. hemophilia treatment centers (HTCs) affiliated with universities. The Inhibitor Prevention Trial is a 48-week randomized phase III trial, in which 66 previously untreated patients (PUPs) with severe hemophilia A will be enrolled. Subjects will include children from 4 months of age up to 4 years of age who have not been previously treated with clotting factor. Once enrolled, subjects who meet all the inclusion and none of the exclusion criteria will be randomized to preemptive weekly Eloctate (rFVIIIFc) vs. weekly Emicizumab (Hemlibra) to prevent inhibitor formation, defined as anti-FVIII >= 0.6 BU. Blood draws will be minimized to 6 timepoints, pre, 4, 12, 24, 36, and 48 weeks, and validated for small volumes, 3.8 cc (¾ tsp) each. The Inhibitor Prevention Trial is considered greater than minimal risk as study drug is given before the first bleed and special inhibitor studies are obtained. (NB: The Inhibitor Prevention Trial (PRO19040140) is linked to the Inhibitor Eradication Trial (PRO19070080), as part of the INHIBIT Clinical Trials Platform, with both trials will be conducted efficiently in the same hemophilia treatment centers (HTCs), with the same MDs, coordinators, visit frequency, blood sampling, and assays.

ELIGIBILITY:
Inclusion Criteria:

1. Male children >= 4 months and up to 4 years of age.
2. Severe hemophilia A (FVIII < 0.01 U/ml).
3. No evidence of an inhibitor i.e. anti-FVIII < 0.6 B.U.
4. No more than 3 FVIII exposures (Factor VIII concentrate, cryoprecipitate, or fresh frozen plasma), including circumcision.

Exclusion Criteria:

1. Acquired hemophilia or any bleeding disorder other than hemophilia A.
2. Treatment with clotting factor or emicizumab previously.
3. Use of an experimental drug(s).
4. Surgery anticipated in the next 48 weeks.
5. Life expectancy less than 5 years.
6. Parent/caretaker unable or unwilling to keep a personal diary of bleeding frequency and study drug treatment, make monthly visits and blood draws at weeks 4, 12, 24, 36, and 48.
7. Other illness, condition or reason in the opinion of the investigator that would make the patient unsuitable for the trial.

Ages: 4 Months to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Arkansas Medical Sciences Childrens Hospital, Little Rock, Arkansas
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - University of Pittsburgh and Hemophilia Center Western PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A biologic specimen and data repository for this trial will be available at the Graduate School of Public Health (GSPH) Data Center repository for investigators who make formal application request and is formally approved by the Coordinating Center (Pitt) and Data Center (GSPH).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year of trial completion.
Access Criteria: Access will be determined by Study Team.

REFERENCES:
- [Background] Ragni MV, George LA; Members of Working Group 1, the NHLBI State of the Science Workshop on factor VIII inhibitors: Generating a national blueprint for future research. The national blueprint for future factor VIII inhibitor clinical trials: NHLBI State of the Science (SOS) Workshop on factor VIII inhibitors. Haemophilia. 2019 Jul;25(4):581-589. doi: 10.1111/hae.13717. PMID 31329364
- [Background] Ebbert PT, Xavier F, Malec LM, Seaman CD, Ragni MV. Observational study of recombinant factor VIII-Fc, rFVIIIFc, in hemophilia A. Thromb Res. 2020 Nov;195:51-54. doi: 10.1016/j.thromres.2020.07.004. Epub 2020 Jul 5. PMID 32653601
- [Background] Bertolet M, Brooks MM, Ragni MV. The design of a Bayesian platform trial to prevent and eradicate inhibitors in patients with hemophilia. Blood Adv. 2020 Nov 10;4(21):5433-5441. doi: 10.1182/bloodadvances.2020002789. PMID 33156923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eloctate
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study closed due to poor enrollment. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eloctate
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 1 [1 to 1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1
Number and Type of Bleeds in the last year [Number; unit: Bleeds] | 0
Prior Circumcision, [Count of Participants; unit: Participants] | 1
Anti-FVIII level > 0.6 BU [Count of Participants; unit: Participants] | 0
Number of FVIII exposures [Number; unit: FVIII exposures] | 0

OUTCOME MEASURES:

1. Primary Outcome: Inhibitor Formation
Description: The proportion developing anti-FVIII inhibitors.
Time Frame: 48 weeks
Population: Only patient was enrolled on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Eloctate
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Bleeding Events
Description: The number of bleeding events:hematoma, joint, central nervous system, other bleeds.
Time Frame: 48 weeks
Population: Only patient was enrolled on study.
Measure: Number; unit: bleeding events
Arm/Group | Eloctate
Number analyzed (Participants) | 1
bleeding events | 1

3. Secondary Outcome: FVIII Trough Level
Description: The FVIII trough activity by chromogenic assay
Time Frame: 48 weeks
Population: specimen collected, discarded with out analysis due to study being close dearly due to low enrollment
Arm/Group | Eloctate
Number analyzed (Participants) | 0

4. Secondary Outcome: Human Leukocyte Antigen (HLA) Haplotype
Description: The number of HLA haplotype variants.
Time Frame: 48 weeks
Population: specimen collected, discarded with out analysis due to study being close dearly due to low enrollment
Arm/Group | Eloctate
Number analyzed (Participants) | 0

5. Secondary Outcome: FVIII Mutation
Description: The number of FVIII mutation variants.
Time Frame: 48 weeks
Population: specimen collected, discarded with out analysis due to study being close dearly due to low enrollment
Arm/Group | Eloctate
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of FVIII Exposures
Description: Number of FVIII exposures,
Time Frame: 48 weeks
Population: Only patient was enrolled on study.
Measure: Number; unit: FVIII exposures
Arm/Group | Eloctate
Number analyzed (Participants) | 1
FVIII exposures | 2

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Adverse events were self-reported.
Arm/Group | Eloctate
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eloctate (N=1)
Joint bleed requiring factor (Blood and lymphatic system disorders) | 1 (1) — Joint bleed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT04303559/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT04303559/ICF_002.pdf